CLINICAL TRIAL: NCT06485934
Title: Development of the Multidimensional Kinesiophobia Scale for the Upper Extremity: A Scale Development Study
Brief Title: Kinesiophobia Scale for the Upper Extremity
Status: Recruiting | Type: Observational
Sponsor: Emre Şenocak (Other)
Responsible Party: Sponsor-Investigator, Emre Şenocak, Research Assistant, Karadeniz Technical University
Organization: Karadeniz Technical University (Other)
Other Study IDs: 2024/74
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Shoulder Injuries
Keywords: Kinesiophobia; Shoulder; Development of Scale
MeSH Terms: conditions — Shoulder Injuries; Kinesiophobia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational Group: All of the outcomes will be applied to patients who come to the outpatient clinic due to shoulder problems. Then, 1 week later, participants will be recalled to apply the multidimensional kinesiophobia scale a second time.

SUMMARY:
Questionnaires/scales used to evaluate kinesiophobia in the literature are limited and are not specific to the upper extremity in existing scales. For this reason, the primary purpose and subject of the study is to develop a multi-factor kinesiophobia scale specific to shoulder problems.

The study is an observational research. Participants will be interviewed twice in total. All primary and secondary outcomes will be assessed at the first meeting. The second come will be performed within 5-7 days after the first assessment. In the second come, only the new kinesiophobia scale that is intended to be developed will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Tampa Kinesiophobia Score >37 points
* Presence of traumatological, orthopedic and rheumatological pathology in the upper extremity
* Mini-Mental State Examination score >24 points

Exclusion Criteria:

* Malignancy,
* Psychiatric drug use,
* Use of painkillers during evaluation periods,
* Those who received physiotherapy before the study (last 6 months),
* Those whose education level is below secondary school level,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Traumatological, orthopedic and rheumatological pathologies that cause fear of movement in the upper extremity
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Multidimensional Kinesiophobia Scale (To be developed) | Baseline of the study
  It is desired to be developed to evaluate the fear of movement that occurs due to upper extremity injuries.
Multidimensional Kinesiophobia Scale (To be developed) | 5-7 days after baseline assessment
  It is desired to be developed to evaluate the fear of movement that occurs due to upper extremity injuries.

SECONDARY OUTCOMES:
Visual Analog Scale | Baseline of the study
  Assesses pain severity. It scores between 0-10 points. A high score indicates high pain intensity.
Tampa Kinesiophobia Scale | Baseline of the study
  It consists of 17 items. Assesses the fear of movement. Total score is 68 points. A high score indicates high fear.
Demographic Data Form | Baseline of the study
  This form was created by researchers and it consist of personal informations such as gender, marital status, education, age, body mass index, dominant and affected extremity, name of pathology,

CONTACTS AND LOCATIONS:
Overall Officials: Abdurrahman Tanhan, PhD, Study Chair — Bitlis Eren University; Zeynep Hoşbay, Associate Professor, Study Chair — Biruni University
Locations (1):
- Clinic of İstanbul Hand-Microsurgery Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided